CLINICAL TRIAL: NCT02272868
Title: Fecal Microbial Transplant in Pediatric Crohn's Disease: A Double Blind Placebo Control Study
Brief Title: Fecal Microbial Transplant in Pediatric Crohn's Disease
Acronym: FMTCD
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, David Suskind, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15262
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fecal microbiome transplant (Experimental): Pretransplant(Rifaximin 400mg tid x 10 days + omeprazole 20 mg night before transplant and day of transplant + miralax 17g tid x 2 days) + Fecal Microbial Transplant
  Interventions: Biological: Fecal Microbial transplant; Drug: rifaximin+omeprazole+miralax
- Normal saline (Placebo Comparator): Pretransplant(Rifaximin 400mg tid x 10 days + omeprazole 20 mg night before transplant and day of transplant + miralax 17g tid x 2 days) + Normal saline
  Interventions: Drug: Normal Saline; Drug: rifaximin+omeprazole+miralax

INTERVENTIONS:
Biological: Fecal Microbial transplant — Pretransplant regimen(rifaxamin+omeprazole+miralax) + Donor feces transplant
  Arms: Fecal microbiome transplant
Drug: Normal Saline — Pretransplant regimen(rifaximin+omeprazole+miralax) +Normal Saline
  Arms: Normal saline
Drug: rifaximin+omeprazole+miralax

SUMMARY:
This is a double blind placebo control trial of fecal microbial transplantation for active Crohn's disease in patients 12 to 21 years of age.

DETAILED DESCRIPTION:
Thirty-two patients with mild to moderate active Crohn's Disease (PCDAI 15-45) aged 12-21 will be enrolled in this study. Patients will be randomized into pre-treatment conditioning + FMT versus pre-treatment conditioning + placebo.

Pre transplant conditioning will include rifaximin (400mg PO three times a day x 10 days prior to transplant), MiraLAX cleanout (2 days prior to cleanout), and omeprazole (day prior and day of transplant). Study subjects will have a nasogastric (NG) tube placed on the day of the transplant after which either donor stool or normal saline (placebo) will be infused via the tube. A designated clinician will do the transplants and keep the subject blinded to the treatment group. A different designated clinician, blinded to the treatment group of the subject, will do the follow-up telephone calls and visits.

Study subjects will have telephone follow up 2 days and at 2, 6 and 12 weeks post transplant they will be seen in clinic. The PCDAI will be completed at all the study visits (excluding the phone call). Additionally, the physcian's global assessment will be documented at each study visit (excluding the phone call). The global assessment will be reported as quiescent, mild, moderate or severe.

Study subject recipients/guardian will be provided diary cards from initiation of rifaximin to 12 weeks post transplant to record AEs, and these will be reviewed at every follow-up encounter. The diary card will include duration of event, intensity of event, and medications or actions taken for the event.

Individuals who received placebo treatment will be offered FMT at termination of study. These patients will then be followed at week 2, 6 and 12 post transplant in the CRC. Donor stool will be saved in the Clinical Research Lab at the initial baseline visit. This stool will be used for the FMT for these individuals.

Randomization The study participants will be randomized using the RedCap database. All study related information will be stored in RedCap for this study. Participant data for the study will be stored electronically in the REDCap platform. The REDCap platform is managed by the Institute for Clinical and Translational Science at the University of Washington. Only IRB approved research team members will have access to the REDCap data platform. Each team members will be granted access to the REDCap data system through a secure login.The information about each participant will be de-identified using a unique study code. The randomization will be set for 16 participants to receive the FMT and 16 participants to receive placebo. For the individuals that receive the placebo, they will have the option to receive the FMT upon completion of the study. The physician that completes the FMT will be the only individual on the study team that is unblinded to the randomization.

Study Procedures:

Screening The screening visit will take place in the Gastroenterology Outpatient Clinic at the Seattle Children's Hospital. At this visit, the subject recipient and donor will review the study in detail with the PI/Research Coordinator. Consent/Assent will be obtained prior to any study activities being performed. The research subject will receive a copy of the Signed Consent/Assent forms for their records. Once Consent/Assent is obtained vital signs including height, weight, blood pressure, heart rate and body temperature will be obtained for the FMT recipient only. Additionally, a physical exam and patient history including the PCDAI, Paris classification and PGA will be completed for the recipient. The FMT donor will complete a lifestyle questionnaire and the physician will review their medical history. Finally, all labs will be completed for the recipient and donor to determine eligibility. The screening labs include both blood and stool tests for both the recipient and donor. Additionally, for FMT recipients, urine will be collected for females of child bearing age for a urine pregnancy test. Some of the stool from the stool recipient will be sent to the University of Washington for microbiome analysis and storage. These samples will be de-identified and labeled with a unique study code and visit number. Consent for storage will be part of the Informed Consent process.

Baseline Once all screening activities are complete and it has been determined that each subject meets all of the inclusion criteria and none of the exclusion criteria the subjects will return to the Pediatric Clinical Research Center at Seattle Children's Hospital to receive or provide the stool/saline transplant. The maximum amount of time that will elapse from donor screening to procurement of stool for transplant (screening to baseline) will be less than 4 weeks.

All FMT/placebo donors will provide a stool sample at this visit regardless of what group the recipient was randomized to (they will not be informed of this information).This is the baseline visit. Prior to this visit, the FMT/placebo recipient will be randomized to a group from the RedCap database. Only the transplant physician will know which group the participant was randomized to. Prior to this visit ALL recipients will take Rifaximin for 10 days (400 mg 3 times/day) prior to the baseline visit. All study recipients will also receive 20 mg Omeprazole the day prior and on the morning of the procedure. The study recipient will also have MiraLAX, 3 times a day for 2 days with the last dose at 5 pm on the evening prior to the PCRC visit. Stool transplant recipient will have stool collected for microbiome analysis at this visit. At this visit, fresh stool from the FMT donor will be obtained. A fresh sample will be defined as being less than 6 hours old. The stool weight will need to be approximately 30 grams. If the child is randomized to the placebo group, the fresh stool sample will be stored in a freezer at -80 °C. At the end of the 12 week period, children that received placebo will be eligible to receive the FMT. At this time, the donor stool will be thawed and processed according to guidelines below for the FMT. The FMT/placebo recipient will arrive fasting to this visit (this means nothing to eat or drink after midnight prior to FMT). Vital signs and a physical exam will be completed at the baseline visit for the study recipient. Additionally, a urine pregnancy test will be completed for all females in the study of child bearing potential (FMT/placebo recipients only). If the test is positive, they will be terminated from the study. After the vital signs are collected and the urine pregnancy test has been completed, a nasogastric tube will be placed for the FMT/placebo recipient. Placement of this tube will be confirmed by abdominal x-ray. The stool from the donor will be placed into a blender and 90 ml of the final suspension will be infused over a 3 minute period through the nasogastric tube. The nasogastric tube will then be flushed with 15 ml of normal saline over 1 minute. After 15 minutes, the nasogastric tube will be removed . The FMT/placebo recipient will be able to be discharged from the CRC after 30 minutes from the stool transplant assuming that their vital signs are stable. The FMT/placebo recipient will resume normal activity after the above procedure. The AE diary and a thermometer for measuring temperature will be given to the subject by the coordinator prior to the discharge. Some of the stool from the FMT donor will be sent to the University of Washington for microbiome analysis and storage. Each of these samples will be de-identified and labeled with a unique study code and consent for storage will be part of the IC process. If the subject is randomized to the placebo arm, all study procedures above will still take place,however, they will receive 90 ml of normal saline instead of donor feces, followed by 15 ml of a normal saline flush. The fresh stool from the stool donor will be stored frozen in the Clinical Research Center (CRC) Lab. The stool from the donor that is stored in the CRC lab will be used for the individuals that initially received placebo. For each group, the syringe will be covered so no one can identify what they are receiving. One clinician will be designated to complete the Fecal transplant. This clinician will not complete any of the follow up visits. After the baseline visit, the stool donors participation will be complete.

Donor stool preparation for FMT

1. Perform hand hygiene and don gloves, a gown, a mask, and an eye shield before stool preparation.
2. Stool should be prepared in a dedicated room in the outpatient procedure area with a dedicated blender, 0.9% saline, and large syringes.
3. Timing of stool collection should be as close to fecal transplant time as possible, and should not be more than 6 hours before the procedure time. If frozen beforehand, please thaw for 1 hour prior to processing.
4. Select stool specimen, preferably a soft one. Add 100-200 mL preservative-free 0.9% saline to 30-70 grams of stool for processing in a conventional, household blender to create a homogenized, liquid slurry.
5. Use the low setting on the blender and blend the stool sample for 2 to 4 minutes until sample is smooth and homogeneous.
6. Strain slurry through a gauze mesh barrier to remove large particulate matter remaining in the slurry. Final prepared stool should be of a smooth consistency.

For Universal Donor Stool Preparation we follow the above preparation and then amended thereafter with sterile pharmaceutical grade glycerol (Sigma, St Louis, MO) to a final concentration of 10 % , and stored frozen at - 80 ° C . The stool suspension will be divided into 90ml aliquots. Each 90 ml aliquot will be use separately. Thawing will be done over 2 - 4 h in an ice bath before the FMT procedure. 9 For universal donor screen the same protocol as for non-universal donor screen will be followed, including the aforementioned donor inclusion and exclusion criteria and screening labs.

Day 2 and Week 24 A telephone interview will occur by a study physician to assure that the study subject recipient is clinically doing well. Any adverse events will be documented at this time. The study physician that completes this call will NOT be the same physician that completed the transplant.

Week 2, week 6 and week 12 Study subjects will return to the Pediatric Clinical Research Center for clinical follow up at approximately 2, 6 and 12 weeks from the day of the FMT/placebo. At each of these visits vital signs including height, weight, blood pressure, heart rate, respiratory rate and body temperature will be obtained. Additionally, a physical exam and the PCDAI and the PGA will be completed. A review of the subjects AE diary will also occur at each of these visits. We will collect blood and stool from the FMT/placebo recipient at each of these visits. Some of the stool from the FMT/placebo recipient will be sent to the University of Washington for microbiome analysis and storage at each visit. Each of these samples will be de-identified and labeled with a unique study code and consent for storage will be part of the IC process.

ELIGIBILITY:
Inclusion criteria for Stool Recipient :Children and adolescents twelve to twenty one years old, Diagnosis of Crohn's disease made by a primary gastroenterologist based upon history, physical exam, laboratory/radiological studies and gastrointestinal histology; Mild or moderate disease activity based upon PCDAI score (15-45); Parent/guardian and child must be able to comprehend the consent and assent in English; Parent/guardian and participant must be able to attend study visits at baseline, and weeks +2, +6, +12.; Patient must not have medication changes for his/her inflammatory bowel disease medications for at least 1 months prior to enrollment.;Stool donor available from family member; Patient agreeable to nasogastric tube placement

Exclusion Criteria for Stool Recipient: PCDAI <15 or PCDAI >45; Active or history of intraabdominal abscess, perianal abscess, perianal fistula, intraabdominal fistula, stricturing Crohn's disease; Other serious medical conditions such as neurological, liver, kidney, autoimmune or systemic disease; recipients allergic to any product used in the study, including rifaximin, omeprazole and MiraLAX; Pregnant or nursing subjects will be excluded as transplant recipients.;Female recipients of child-bearing potential will abstinent or willing to use adequate birth control from screening until the end of the study. ; Patients who cannot tolerate NG tube placement, such as those with recent surgery or trauma to the nares will be excluded; Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data;

Stool donor inclusion criteria: Family member of child participant with IBD over the age of 18 or Universal Donor known to the PI/co-PI; Willing and able to donate a stool sample

Exclusion criteria for Stool donors: High risk behaviors as outlined in the American Association of Blood Banks Donor History Questionnaire; confirmed lab positivity for: Hepatitis A(IgM),Hepatitis B (serum antigen, core antibody), Hepatitis C (IgG or IgM), HIV 1-2 (PCR), Syphilis (IgG and IgM), EBV(IgM), CMV(IgM) ; Stool sample positive for: c. difficile, salmonella species, shigella species, campylobacter species, Aeromonas hydrophila, yersinia, vibrio parahaemolyticus, vibrio cholerae, e. coli H-0157, H. Pylori, listeria, protozoa, trophozoites and cysts, helminths and ova; Antibiotic use during the 3 months prior to the stool transplant; Diagnosis of IBD, polyposis syndrome, gastrointestinal malignancy in stool donor; Currently on major immunosuppressant medications for example, exogenous glucocorticoids, biological agents, and calcineurin inhibitors; Use of investigational product(s) during the month prior to donation or expected use from screening to donation; Metabolic syndrome or history of bariatric surgery; Diarrheal illness or blood in stool within the month prior to screening; Pregnancy; Malignancy or use of systemic chemotherapy ; Autoimmune disease; Chronic pain syndrome; Atopic disease;Recent ingestion of a potential allergen where recipient has a known allergy to the agent; Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or the quality of the data.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Pediatric Crohn's Disease Activity Index | 12 weeks
  Clinical disease activity index in Crohn's disease

CONTACTS AND LOCATIONS:
Overall Officials: David Suskind, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- See also: Physician Link — http://www.seattlechildrens.org/medical-staff/David-L-Suskind/